CLINICAL TRIAL: NCT07379723
Title: Feasibility Pilot Study of a Brief Intervention in Functional Cognitive Disorder
Brief Title: Brief Intervention for FCD: A Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRAS Reference: 354504
Record Dates: First submitted 2026-01-14; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Functional Cognitive Disorder
Keywords: Functional Cognitive Disorder; Brief Interventions; Feasibility; Pilot; Attention Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: Brief psychological intervention including attention training

INTERVENTIONS:
Behavioral: Brief psychological intervention including attention training — Brief psychological intervention including attention training

SUMMARY:
The goal of this study is to learn if a single session intervention for people with Functional Cognitive Disorder (FCD) is feasible and acceptable. The main questions it aims to answer are:

What is the impact of a single session intervention on FCD symptoms, functional impairment, and quality of life in people with FCD?

What is the feasibility and acceptability of piloting a single session intervention for people with FCD.

Participants will:

* Complete questionnaires about cognitive concerns, anxiety, depression, functional impairment and quality of life
* Visit the clinic for a single session intervention including practicing the Attention Training Technique (ATT)
* Complete 2 telephone calls with a researcher to discuss their use of the intervention and to complete the same questionnaires from their clinic visit, and a questionnaire about their experience of the study and intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 or below
* Meet criteria for diagnosis of FCD (criteria include normal MRI results with no neurological diagnosis, and symptoms that are not explained by any other medical condition, performance at routine pre-baseline neuropsychological assessment within the service)
* Not taking part in any other intervention study or trial

Exclusion Criteria:

* Aged above 65 years
* Lack capacity to consent
* MRI results not in normal range
* Neurological diagnosis
* Indication of severe low mood or depression (from clinical interview, routine measures)
* Taking part in any other intervention study or trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Participant recruitment, feasibility and retention from baseline to follow-up | From enrollment to follow-up 6 weeks post-intervention.
  • Number of participants recruited and retention rate (number and percentage of participants completing post-intervention measures) will be recorded.

SECONDARY OUTCOMES:
Acceptability of the study intervention at follow-up | Post-intervention follow-up at 6 weeks.
  • At follow-up, participants will complete a questionnaire to collect information on acceptability of the study and intervention (Theoretical framework of acceptability [TFA] questionnaire; Sekhon et al., 2022).
Change in symptoms of depression from enrolment to post-intervention follow-up | At enrolment and at follow-up 6 weeks post-intervention
  Participants will complete questionnaire at enrolment and at follow-up post-intervention:
  • Patient Health Questionnaire 9 (PHQ-9) (Kroenke et al., 2001)
Change in symptoms of anxiety from enrolment to post-intervention follow-up | At enrolment and at follow-up 6 weeks post-intervention
  Participants will complete questionnaire at enrolment and at follow-up post-intervention:
  • Generalised Anxiety Disorder 7 questionnaire (GAD- 7) (Spitzer et al., 2006)
Change in functional impairment from enrolment to post-intervention follow-up | At enrolment and at follow-up 6 weeks post-intervention
  Participants will complete questionnaire at enrolment and at follow-up post-intervention:
  • Work and Social Adjustment Scale (WSAS) (Mundt et al., 2002)
Change in quality of life from enrolment to post-intervention follow-up | At enrolment and at follow-up 6 weeks post-intervention
  Participants will complete questionnaire at enrolment and at follow-up post-intervention:
  • EuroQol 5-Dimension 5-Level (EQ-5D-5L)(Herdman et al., 2011)
Change in self-reported cognitive symptoms from enrolment to post-intervention follow-up | At enrolment and at follow-up 6 weeks post-intervention
  Participants will complete questionnaire at enrolment and at follow-up post-intervention:
  • The Cognitive Failures Questionnaire 2.0(Goodhew & Edwards, 2024).

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No